CLINICAL TRIAL: NCT00273026
Title: An Open-label, Multi-centre, Randomized, Parallel Group Clinical Effectiveness Study to Determine the Level of Asthma Control in Adolescent and Adult Patients With ADVAIR Versus Usual Care for 24 Weeks.
Brief Title: Study In Asthma Control
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SFA103081
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Asthma
Keywords: Asthma Advair
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination

INTERVENTIONS:
Drug: salmeterol xinafoate/fluticasone propionate

SUMMARY:
This study will compare patients treated with a marketed medication and those who continue with their usual care to assess the proportion of patients achieving well controlled asthma after 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* documented clinical history of asthma and receiving regular maintenance therapy.

Exclusion Criteria:

* Using oral/parenteral or depot corticosteroids within 12 weeks of visit 1.
* History of heavy smoking or substance abuse.
* Females who are pregnant or lactating.
* Required emergency room treatment for their asthma 12 weeks prior to Visit 1.
* Serious, uncontrolled, systemic disease that may make study participation unsafe or inappropriate in the opinion of the physician.
* Other medical criteria will be evaluated at the screening visit.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 680
Dates: Start 2004-11-08; Study Completion 2006-03-28 (Actual)

PRIMARY OUTCOMES:
Percentage of patients achieving well-controlled asthma at the end of the treatment period.

SECONDARY OUTCOMES:
Percentage of patients achieving total asthma control as defined by the Canadian Asthma consensus guidelines at the end of the treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (78):
- Canada (78):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Abbotsford, British Columbia
  - GSK Investigational Site, Burnaby, British Columbia
  - GSK Investigational Site, Chilliwack, British Columbia
  - GSK Investigational Site, Coquitlam, British Columbia
  - GSK Investigational Site, Delta, British Columbia
  - GSK Investigational Site, Kamloops, British Columbia
  - GSK Investigational Site, Kelowna, British Columbia
  - GSK Investigational Site, Maple Ridge, British Columbia
  - GSK Investigational Site, Penticton, British Columbia
  - GSK Investigational Site, Richmond, British Columbia
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Brandon, Manitoba
  - GSK Investigational Site, Steinbach, Manitoba
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Moncton, New Brunswick
  - GSK Investigational Site, Rothesay, New Brunswick
  - GSK Investigational Site, Bay Roberts, Newfoundland and Labrador
  - GSK Investigational Site, Holyrood, Newfoundland and Labrador
  - GSK Investigational Site, Mount Pearl, Newfoundland and Labrador
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Bridgewater, Nova Scotia
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Upper Tantallon, Nova Scotia
  - GSK Investigational Site, Ajax, Ontario
  - GSK Investigational Site, Barrie, Ontario
  - GSK Investigational Site, Bolton, Ontario
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Brantford, Ontario
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, Fort Erie, Ontario
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Kanata, Ontario
  - GSK Investigational Site, Kingston, Ontario
  - GSK Investigational Site, Kitchener, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Newmarket, Ontario
  - GSK Investigational Site, Niagara Falls, Ontario
  - GSK Investigational Site, North Bay, Ontario
  - GSK Investigational Site, North York, Ontario
  - GSK Investigational Site, Oshawa, Ontario
  - GSK Investigational Site, Peterborough, Ontario
  - GSK Investigational Site, Prescott, Ontario
  - GSK Investigational Site, Renfrew, Ontario
  - GSK Investigational Site, Richmond Hill, Ontario
  - GSK Investigational Site, Saint Catherines, Ontario
  - GSK Investigational Site, Scarborough Village, Ontario
  - GSK Investigational Site, Thornhill, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Trenton, Ontario
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Brossard, Quebec
  - GSK Investigational Site, Charlesbourg, Quebec
  - GSK Investigational Site, Châteauguay, Quebec
  - GSK Investigational Site, Chicoutimi, Quebec
  - GSK Investigational Site, Contrecoeur, Quebec
  - GSK Investigational Site, Courcelette, Quebec
  - GSK Investigational Site, Cowansville, Quebec
  - GSK Investigational Site, LaSalle, Quebec
  - GSK Investigational Site, LeGardeur, Quebec
  - GSK Investigational Site, Longueuil, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Princeville, Quebec
  - GSK Investigational Site, Saine-Eustache, Quebec
  - GSK Investigational Site, Saint Romuald, Quebec
  - GSK Investigational Site, Sainte Jerome, Quebec
  - GSK Investigational Site, Sainte-Catherine, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
  - GSK Investigational Site, St-Bruno, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
  - GSK Investigational Site, Ville Lasalle, Quebec
  - GSK Investigational Site, Regina, Saskatchewan
  - GSK Investigational Site, Saskatoon, Saskatchewan
  - GSK Investigational Site, Québec